CLINICAL TRIAL: NCT03102905
Title: Prevalence of Replication of Human Herpes Virus 6 (HHV6) in Blood and Skin During Exanthemia, in Patients With Hemopathy. Is There a Correlation With the Etiology of the Exanthema?
Acronym: REPLIPO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2016_843_0017
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-03

CONDITIONS: HHV6; Exanthema; Hemopathy
MeSH Terms: conditions — Exanthema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measurement of the prevalence of the positivity of cutaneous HHV6 quantitative PCR in the cohort studied. — To evaluate the prevalence of the positivity of HHV6 PCR in the skin, during the exanthema in patients hospitalized for haemopathy.

SUMMARY:
To look for the replication of HHV6 by PCR in the skin, in these patients with haemopathies presenting an exanthema. This will make it possible to evaluate the prevalence of the positivity of this PCR in the skin. Then the investigator can investigate whether there is an association between the positivity of HHV6 PCR in the blood and / or skin and the viral etiology of the exanthema. If this association exists, it will make it possible to improve the diagnosis in the context of the exanthema and thus to improve the therapeutic management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Supported for any type of hemopathy.
* Allograft, autografted or ungrafted haematopoietic stem cells
* Having presented an exanthema during hospitalization, for which a cutaneous biopsy had been performed
* Having had a blood test of the HHV6 virus by PCR at least within the previous 40 days or following the rash.
* Age greater than or equal to 18 years
* Patient informed of the protocol by post, not having refused within one month of sending the said courier.

Exclusion Criteria:

* Patient who refused the search.
* Patient whose HHV6 PCR in the blood was carried out at a distance of more than 40 days from the skin biopsy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient hospitalized in the Clinical Hematology and Cellular Therapy department of the CHU Amiens-Picardie between 01/01/2011 and 31/01/2016
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2017-06-13 (Estimated); Study Completion 2017-06-13 (Estimated)

PRIMARY OUTCOMES:
Measurement of the prevalence of the positivity of cutaneous HHV6 quantitative PCR in the cohort studied. | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France